CLINICAL TRIAL: NCT01445236
Title: Pilot Study of Immunosuppression Drug Weaning in Liver Recipients Exhibiting Biomarkers of High Likelihood of Tolerance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Alberto Sanchez-Fueyo, Director IDIBAPS Transplant Immunology Laboratory, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Weaning-Biomarkers
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Liver Transplantation
Keywords: Operational tolerance; Biomarkers; Liver Transplantation
MeSH Terms: interventions — Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Weaning patients (Experimental)
  Interventions: Other: Immunosuppresion withdrawal

INTERVENTIONS:
Other: Immunosuppresion withdrawal — Gradual discontinuation of all immunosuppressive drugs.
  Other Names: Cyclosporine A; Tacrolimus

SUMMARY:
Immunosuppressive drugs can be successfully withdrawn in a fraction of liver transplant patients. Specific peripheral blood gene expression markers can be employed to select patients with a high likelihood of being tolerant. In the current study the investigators propose to conduct a pilot non-randomized prospective study in which gradual weaning of immunosuppressive drugs will be offered to liver recipients exhibiting a favorable peripheral blood gene expression profile.

DETAILED DESCRIPTION:
HYPOTHESIS We hypothesize that liver recipients exhibiting either specific gene expression and/or cell phenotypic markers in peripheral blood will be successfully weaned from all immunosuppressive drugs.

OBJECTIVE Evaluate the applicability of a set of non-invasive biomarkers in the identification of liver transplant recipients who can successfully discontinue all immunosuppressive therapy.

METODOLOGY

1. Immunosuppression drug weaning: according to the clinical protocol approved, all patients will undergo liver biopsy before entry. Patients will be visited every 4 weeks, and immunosuppressive drugs will be gradually discontinued with the aim of achieving 50% decrease in drug dosages by month 3, and complete withdrawal by month 6 after initiation of the study. Following drug discontinuation, patients will continue to be followed every month until month 12 after initiation of the study. Liver function tests will be obtained at every clinical follow-up visit.
2. Management of liver function test alterations: a) Increases in liver function tests below 2-fold normal levels for AST/ALT/GGT or 1.5-fold normal levels for ALP will result in no further decreases in drug dosages, and performance of new liver function tests in 14 days. Worsening or persistence of liver function test alterations will constitute indication for liver biopsy. b) Increases in liver function tests beyond 2-fold normal levels for AST/ALT/GGT or1.5-fold normal levels for ALP.
3. Diagnosis of liver graft rejection: will be based on the finding of 2 out of 3 of the following histological criteria: portal inflammation, injury to bile duct epithelium, and endothelitis. The finding of a mixed portal/loblular lymphocytic infiltrate not attributable to any other cause and responding to an increase in immunosuppressive drug doses will also be considered as a rejection.
4. Management of rejection episodes: patients presenting with mild to moderate acute rejection will be treated with 20 mg of prednisone in decreasing doses within 4 to 6 weeks. Patients with severe acute rejection will be admitted to hospital and treated with high dose IV prednisone (500-1000mg/day) during 3 day and thereafter oral prednisone at decreasing dose according to evolution of liver function tests. In every case patients will return to previous immunosuppressive dose enough to maintained normal or near normal liver function test.

SAMPLE SIZE According to our data, the success rate of an immunosuppression withdrawal strategy in stable liver transplant recipients transplanted for more than 3 year is 42% (these patients are consider as operationally tolerants). Our hypothesis is that with the use of biomarkers to identify potential tolerant patients the investigators will be able to increase the success rate of this strategy up to 78%. In order to achieve this success rate the sample size needed in this study is 25 patients (power 80% and significance of 95%).

ELIGIBILITY:
Inclusion Criteria:

1. Liver transplant recipients with at least 3 years of post-operative follow-up in whom gene expression pattern changed from non-tolerant to tolerant under sirolimus treatment.
2. Feasibility of performing very frequent (every 2-3 weeks) clinical follow-up visits.
3. No history of graft rejection during the previous 12 months.
4. Basal liver biopsy without signs of rejection
5. Stability of liver graft function, defined as: a) normal liver function tests (AST, ALT, ALP, GGT) during at least 6 months; or alternatively b) minor alterations in liver function tests that have not changed over the previous 6 months (AST/ALT < 2 fold normal levels; ALP < 1.5 fold normal levels; GGT < 2 fold normal levels; bilirubin < 2 mg/dL).
6. Presence of peripheral blood biomarkers of high likelihood of tolerance as defined by: a) transcriptional pattern associated with tolerance regardless of the basal immunosuppressive regimen; and/or b) 2-fold increase in Treg frequency in patients who have discontinued calcineurin inhibitors in the 12 months prior to inclusion.
7. Signature of informed consent.

Exclusion Criteria:

1. Requirement of immunosuppressive treatment for an indication different to liver transplantation.
2. Documented human immunodeficiency virus (HIV) infection.
3. Liver-Kidney transplant recipients.
4. History of liver autoimmune disease (autoimmune hepatitis, primary liver cirrhosis, primary sclerosing cholangitis)
5. Active hepatitis C virus infection as defined by positive serum HCV-RNA.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients developing operational tolerance | 12 months after complete withdrawal of all immunosuppressive drugs

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sanchez-Fueyo, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain